CLINICAL TRIAL: NCT03129880
Title: Voice-related Outcomes in Response to Intensive Versus Traditional Therapy Programs
Brief Title: Intensive Versus Traditional Voice Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0763; A539772 (Other: UW Madison); SMPH/SURGERY/SPEECH (Other: UW Madison); Protocol Version 12/2/2020 (Other: Minimal Risk IRB (Health Sciences), UW Madison)
Record Dates: First submitted 2017-04-18; First posted 2017-04-26 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Dysphonia
Keywords: Voice disorder; Hoarseness; Phonation Disorders; Speech Disorders
MeSH Terms: conditions — Dysphonia; Voice Disorders; Hoarseness; Speech Disorders

STUDY DESIGN:
Intervention Model Description: For purposes of this study participants will be randomized into one of the following two groups:
  4-6 weekly standard of care therapy sessions, once a week, for a maximum of six weeks 4-6 standard of care therapy sessions in one day Standard of care treatment may continue past patient enrollment in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weekly Voice Therapy (Placebo Comparator): Participants are randomized to receiving weekly voice therapy sessions
  Interventions: Behavioral: Weekly Voice Therapy
- Intensive Voice Therapy (Active Comparator): Participants are randomized to receiving multiple sessions of voice therapy in one day
  Interventions: Behavioral: Intensive Voice Therapy

INTERVENTIONS:
Behavioral: Weekly Voice Therapy — Participants will be randomized to receive weekly voice therapy
  Arms: Weekly Voice Therapy
Behavioral: Intensive Voice Therapy — Participants will be randomized to receive multiple sessions of voice therapy in one day.
  Arms: Intensive Voice Therapy

SUMMARY:
The purpose of this study is to determine if there are differences in treatment outcomes between traditional voice therapy, performed weekly for a maximum of 6 weeks versus intensive voice therapy, consisting of 4-6 therapy sessions performed within one day.

DETAILED DESCRIPTION:
The goal of voice therapy is optimal long-term vocal quality and communication function with minimal recurrence. Traditional voice therapy for dysphonia typically consists of one to two therapy sessions each week with a single clinician for about 8 weeks. Another approach of voice therapy is intensive short-term therapy also known as "boot camp." This approach, borrows from the disciplines of neurobiology, exercise physiology, motor learning, and psychotherapy which describe desirable learning and behavior changes influenced by practice that involves high-intensity overload, variability, and specificity of training. A few studies have showed that "Boot Camp" model of intensive therapy resulted in comparable gains in voice quality and vibratory mechanics and may promote better patient satisfaction and attendance.

While such findings support the notion that intensive voice therapy may enhance voice therapy outcomes, no study to date has examined patient response to the "Boot Camp" approach to voice therapy. The investigators will compare the outcomes of traditional, weekly voice therapy and intensive voice therapy with multiple sessions in one day.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a Voice disorder
* Diagnosed with benign vocal fold lesions and/or hyper-function
* First/primary propose treatment modality is voice therapy
* Patients who are appropriate for either standard of care treatment modality (traditional or intensive voice therapy)
* Willingness to participate in either standard of care treatment modality
* All races
* Males and females
* English speaking

Exclusion Criteria:

* Younger than 18
* Inability or unwillingness to participate in one of the standard of care treatment modalities
* Laryngeal Surgery or procedures during course of study
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-03-13 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Self-efficacy and readiness scale Changes | Baseline compared to Immediately post voice therapy
  Pre to Post difference in participant's self-efficacy for voice practice and healthy voice technique between therapy groups and within subsets of subjects - readiness ruler of 0 (not at all) to 10 (extremely)
Self-efficacy and readiness scale Change | Baseline compared to 12 weeks post voice therapy
  Pre to Post difference in participant's self-efficacy for voice practice and healthy voice technique between therapy groups and within subsets of subjects - readiness ruler of 0 (not at all) to 10 (extremely)

CONTACTS AND LOCATIONS:
Overall Officials: Emerald J Doll, MS, CCC-SLP, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison Voice and Swallow Clinic, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No